CLINICAL TRIAL: NCT06329089
Title: RENATA Study: Reoperative Sentinel Lymph Node Biopsy in Patients With Recurrent Ipsilateral Breast Cancer and Prior Axillary Surgical Techniques and Approaches
Brief Title: Reoperative Sentinel Lymph Node Biopsy in Patients With Recurrent Ipsilateral Breast Cancer
Acronym: RENATA
Status: Recruiting | Type: Observational
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Other Study IDs: HCB/2023/0840
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Recurrent Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Recurrent ipsilateral breast cancer: Recurrent ipsilateral breast cancer refers to the return of breast cancer in the same breast where it originally developed or was treated.
  Interventions: Procedure: Reoperative Sentinel Lymph Node Biopsy

INTERVENTIONS:
Procedure: Reoperative Sentinel Lymph Node Biopsy — Reoperative sentinel lymph node biopsy refers to a surgical procedure performed when there is a need to re-examine the sentinel lymph nodes (SLNs) in patients who have previously undergone breast cancer surgery. The sentinel lymph nodes are the first lymph nodes to which cancer cells are likely to spread from the primary tumor. During the procedure, the surgeon locates and removes the previously identified sentinel lymph nodes using techniques such as lymphatic mapping and injection of a radiotracer or dye. The removed lymph nodes are then examined by a pathologist to determine if there is any evidence of cancer spread.

SUMMARY:
The goal of this observational study is to assess the effectiveness of sentinel lymph node biopsy as a treatment approach for patients with recurrent breast cancer on the same side as previous surgeries. The main questions it aims to answer are:

* What is the rate of identification of the sentinel lymph node, and how does it vary among patients with different histories of axillary surgeries?
* How can we describe and understand the drainage pathways, including those from the armpit on the same side as the cancer, the area near the breastbone, and the opposite armpit?

Participants will undergo sentinel lymph node biopsy as part of their treatment for recurrent breast cancer. They will also receive standard treatments, including surgery and adjuvant therapies as recommended by their healthcare team.

DETAILED DESCRIPTION:
Prospective multicentric collection will be conducted for all patients diagnosed with ipsilateral recurrent breast cancer, who meet the criteria and are eligible for surgery, and who wish to participate in the study. Additional examinations and treatments will be performed according to standard clinical practice. Tests not included in routine practice will not be conducted.

Suspicion of axillary involvement will be ruled out using ultrasound or magnetic resonance imaging, as well as distant metastasis with standard staging studies (bone scintigraphy/computed tomography of the thorax, abdomen, and pelvis).

Lymphatic mapping will be performed according to each hospital's protocol, similar to lymphatic mapping in primary breast cancer. The radiotracer/dye will be injected according to each center's standard practice (peritumoral, intratumoral, intradermal, or periareolar in the quadrant of the tumor) the day before or on the day of surgery by Nuclear Medicine/Radiology. Lymphoscintigraphy will be performed, and the detected sentinel lymph nodes (SLNs) will be marked on the skin with ink/marker. In cases where the SLN is not visualized, a second dose of radiotracer may be administered.

If there is no drainage from the SLN and no prior lymphadenectomy (LA), additional axillary surgery will not be performed. If there is no drainage from the SLN and no prior LA, consideration will be given to performing lymphadenectomy according to each center's protocol.

During surgery, SLNs will be identified using a gamma probe and/or dye, with assistance from the nuclear medicine service. Between one and three SLNs will be removed (whether drainage is in the ipsilateral axilla, internal mammary, or contralateral axilla). They will be sent to Pathology for intraoperative or deferred examination (by One-Step Nucleic Acid Amplification (OSNA) or conventional technique).

If infiltration is found in any of the axillary SLNs (isolated tumor cells, micrometastasis, or macrometastasis), axillary surgery will be completed with a lymphadenectomy including levels I and II of Berg. If infiltration is found in internal mammary SLNs and not in axillary SLNs, irradiation of the internal mammary chain will be performed (recommended dose of 50 Gy), without completing the LA. If contralateral axillary SLNs are affected, further treatment will be decided by consensus in the subsequent treatment committee.

A wound care visit with a specialized breast unit nurse will be scheduled for the week after surgery to assess postoperative complications, and an outpatient consultation with Gynecology will be scheduled for 3 weeks after surgery for further evaluation.

Adjuvant treatment will be administered according to consensus in the hospital's multidisciplinary committee, following standard practice.

Follow-up will be conducted in outpatient consultations with Gynecology/Medical Oncology/Radiation Oncology, with physical examination every 4-6 months, and annual mammography and ultrasound, as per the consensus of the hospital's breast unit. A validated Spanish-language quality of life questionnaire following breast surgery (BREAST-Q) will be administered by Gynecology at 12 months post-surgery, along with evaluation of late postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old with ipsilateral local recurrence of breast cancer with clinical stage cT1-3 cN0 confirmed by histology, with a history of previous axillary surgery (both sentinel lymph node biopsy and lymphadenectomy).

Exclusion Criteria:

* Patients with confirmed axillary metastasis (histology/immunohistochemistry)
* Inflammatory carcinoma
* Patients with suspected or confirmed distant metastasis on staging studies
* Inability to perform the sentinel lymph node biopsy technique: allergy to radiotracer, mobility limitation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises individuals who are over 18 years old and have been diagnosed with ipsilateral local recurrence of breast cancer, confirmed histologically with tumor sizes ranging from clinical stage cT1 to cT3. These patients must have a history of prior axillary surgery, including both sentinel lymph node biopsy and lymphadenectomy.
  Exclusion from the study includes patients with confirmed axillary metastasis, diagnosed inflammatory carcinoma, or suspected or confirmed distant metastasis based on staging studies. Additionally, individuals unable to undergo sentinel lymph node biopsy due to allergies to the radiotracer or mobility limitations are excluded from participation.
Sampling Method: Probability Sample
Enrollment: 97 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Re-Sentinel Lymph node harvesting rate | 12 months
  Calculation of SLN identification rate and analysis of subgroups based on previous axillary surgery.
Drainage pathways description | 12 months
  Describe and study the drainage pathways including the ipsilateral axilla, the internal mammary chain, and the contralateral axilla

SECONDARY OUTCOMES:
Complications rate | 12 months
  Analyze the surgical complications of the axillary, internal mammary, and contralateral axillary SLN technique in patients with previous axillary surgery.
Axillary metastasis rate | 12 months
  Calculate the rate of axillary metastatic infiltration and lymphadenectomy in patients with ipsilateral recurrent breast cancer and axillary negative clinical stage (cN0)
Correlation Between Axillary and Internal Mammary Chain Infiltration | 12 months
  Investigate the relationship between axillary and internal mammary chain infiltration
Quality of life in recurrent breast cancer | 12 months
  Assess the quality of life in patients undergoing re-intervention for ipsilateral recurrent breast cancer using a validated questionnaire (Breast-Q).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No